CLINICAL TRIAL: NCT04935398
Title: Efficacy of Manual Therapy Combined With an Exercise Programme Versus Combined Electrotherapy on Football Players With Adductor Tendinopathy: Randomised Clinical Trial
Brief Title: Efficacy of Manual Therapy Combined With an Exercise Programme VS Combined Electrotherapy on Football Players With Adductor Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica de Ávila (Other)
Responsible Party: Principal Investigator, JORGE VELAZQUEZ SAORNIL, Principal investigator, Universidad Católica de Ávila
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 28/05/2021
Record Dates: First submitted 2021-05-28; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Tenopathy; Lower Limb
Keywords: manual therapy,; electrotherapy,; groin pain and adductors.
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Simple blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual therapy (Experimental): Football players with adductor tendinopathy undergoing treatment consisting of manual therapy and therapeutic exercise.
  Interventions: Other: Physiotherapy
- Electrotherapy (Experimental): Footballers with adductor tendinopathy undergoing electrotherapy treatment
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — The aim is to test two treatment techniques against each other to see how effective they are.

SUMMARY:
Background: Groin pain associated with adductor tendinopathy is the second cause of muscle pathology in a football player (20%), so a good treatment taking into account both internal and external factors that may influence the pathology of our patient, would be the key to an improvement in the symptoms he may have. Material and methods: Firstly, the pain threshold is measured by performing the Copenhagen compression test, and in a palpation at the proximal level of the adductors, the hip joint range (ROM) is measured and the HAGOS questionnaire is passed. Then, a sample of 20 participants (N = 20) is selected and randomly divided into two groups, a control group of 10 participants (n = 10), with a treatment based on electrotherapy combined with an exercise programme; and an experimental group of 10 participants (n = 10) with a treatment based on manual therapy combined with an exercise programme. Finally, they performed all measurements.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 15 and 30 years old.
* Third division and third year national youth football players.
* Males.
* Average of 3 training sessions and 1 match per week.
* Pain when performing the Copenhagen test or Squeeze test for 5 seconds (s).
* Pain on palpation of the proximal insertion of the adductors.

Exclusion Criteria:

* Players over 30 years of age and under 15 years of age.
* Players with previous adductor surgery.
* Players with inguinal hernia.
* Players with signs or symptoms of urinary or genital pathology.
* Players unable to attend study treatment sessions.
* Players on medication during treatment.
* Players who are undergoing other treatment for groin pathology or have had previous treatment of less than one month.

previous treatment of less than one month.

Ages: 15 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Satisfaction assessed by the Visual Analogue Scale | 30 days
  Visual analogue scale that measures the subjective pain of each individual. It is distributed from zero to ten, where zero is the minimum pain reported by the individual and ten is the maximum pain endured.

SECONDARY OUTCOMES:
Range of motion, articular | 30 days
  Observe range of motion, articular
Rate of functionality | 30 days
  Measuring functionality after treatment in adductor tendinopathy

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica de Ávila, Ávila, Spain

IPD SHARING:
Plan to Share IPD: No
In the future, it is planned to share the research study with the rest of the scientific community through a paper submitted to a leading research journal.

REFERENCES:
- [Result] Hopp SJ, Culemann U, Kelm J, Pohlemann T, Pizanis A. Osteitis pubis and adductor tendinopathy in athletes: a novel arthroscopic pubic symphysis curettage and adductor reattachment. Arch Orthop Trauma Surg. 2013 Jul;133(7):1003-9. doi: 10.1007/s00402-013-1777-7. Epub 2013 May 21. PMID 23689650
- [Result] Holmich P, Larsen K, Krogsgaard K, Gluud C. Exercise program for prevention of groin pain in football players: a cluster-randomized trial. Scand J Med Sci Sports. 2010 Dec;20(6):814-21. doi: 10.1111/j.1600-0838.2009.00998.x. PMID 19883386
- [Result] Jansen JA, Mens JM, Backx FJ, Kolfschoten N, Stam HJ. Treatment of longstanding groin pain in athletes: a systematic review. Scand J Med Sci Sports. 2008 Jun;18(3):263-74. doi: 10.1111/j.1600-0838.2008.00790.x. Epub 2008 Apr 6. PMID 18397195
- [Result] Paajanen H, Hermunen H, Karonen J. Pubic magnetic resonance imaging findings in surgically and conservatively treated athletes with osteitis pubis compared to asymptomatic athletes during heavy training. Am J Sports Med. 2008 Jan;36(1):117-21. doi: 10.1177/0363546507305454. Epub 2007 Aug 16. PMID 17702996
- [Result] Crane JD, Ogborn DI, Cupido C, Melov S, Hubbard A, Bourgeois JM, Tarnopolsky MA. Massage therapy attenuates inflammatory signaling after exercise-induced muscle damage. Sci Transl Med. 2012 Feb 1;4(119):119ra13. doi: 10.1126/scitranslmed.3002882. PMID 22301554
- [Result] Sefton JM, Yarar C, Carpenter DM, Berry JW. Physiological and clinical changes after therapeutic massage of the neck and shoulders. Man Ther. 2011 Oct;16(5):487-94. doi: 10.1016/j.math.2011.04.002. Epub 2011 May 12. PMID 21570335
- [Result] Machotka Z, Kumar S, Perraton LG. A systematic review of the literature on the effectiveness of exercise therapy for groin pain in athletes. Sports Med Arthrosc Rehabil Ther Technol. 2009 Mar 31;1(1):5. doi: 10.1186/1758-2555-1-5. PMID 19331695
- [Result] Pauli S, Willemsen P, Declerck K, Chappel R, Vanderveken M. Osteomyelitis pubis versus osteitis pubis: a case presentation and review of the literature. Br J Sports Med. 2002 Feb;36(1):71-3. doi: 10.1136/bjsm.36.1.71. PMID 11867499
- [Result] Weir A, Jansen JA, van de Port IG, Van de Sande HB, Tol JL, Backx FJ. Manual or exercise therapy for long-standing adductor-related groin pain: a randomised controlled clinical trial. Man Ther. 2011 Apr;16(2):148-54. doi: 10.1016/j.math.2010.09.001. Epub 2010 Oct 16. PMID 20952244
- [Result] Moreno-Perez V, Travassos B, Calado A, Gonzalo-Skok O, Del Coso J, Mendez-Villanueva A. Adductor squeeze test and groin injuries in elite football players: A prospective study. Phys Ther Sport. 2019 May;37:54-59. doi: 10.1016/j.ptsp.2019.03.001. Epub 2019 Mar 2. PMID 30856592
- [Result] Serner A, van Eijck CH, Beumer BR, Holmich P, Weir A, de Vos RJ. Study quality on groin injury management remains low: a systematic review on treatment of groin pain in athletes. Br J Sports Med. 2015 Jun;49(12):813. doi: 10.1136/bjsports-2014-094256. Epub 2015 Jan 29. PMID 25633830
- [Result] Short S, Short G, Strack D, Anloague P, Brewster B. A COMBINED TREATMENT APPROACH EMPHASIZING IMPAIRMENT-BASED MANUAL THERAPY AND EXERCISE FOR HIP-RELATED COMPENSATORY INJURY IN ELITE ATHLETES: A CASE SERIES. Int J Sports Phys Ther. 2017 Nov;12(6):994-1010. PMID 29158960
- [Result] Schoberl M, Prantl L, Loose O, Zellner J, Angele P, Zeman F, Spreitzer M, Nerlich M, Krutsch W. Non-surgical treatment of pubic overload and groin pain in amateur football players: a prospective double-blinded randomised controlled study. Knee Surg Sports Traumatol Arthrosc. 2017 Jun;25(6):1958-1966. doi: 10.1007/s00167-017-4423-z. Epub 2017 Jan 16. PMID 28093636